CLINICAL TRIAL: NCT00914875
Title: Kidney Function After Laparoscopic Cholecystectomy and Tramadol Anesthesia Plus Dipyrone or Ketorolac
Brief Title: Kidney Function After Pneumoperitoneum and Analgesia
Status: Completed | Type: Observational
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Clinical Research Ethic Comittee of Botucatu Medical School, Botucatu Medical School
Other Study IDs: upeclin/HC/FMB-Unesp-25
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Last update posted 2009-06-05 (Estimated); Status verified 2009-06

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: kidney function tests; anti-inflammatory agents, non-steroidal; laparoscopic cholecystectomy; adult

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- group tramadol plus ketorolac
- group tramadol plus dypirone

SUMMARY:
double blind study of kidney function of two groups of adult patients submitted to laparoscopic cholecystectomy and analgesia from tramadol associated to dipyrone or ketorolac

DETAILED DESCRIPTION:
Background: The laparoscopic cholecystectomy (LC) reduces surgical trauma and hospital stay but requires effective and safe postoperative analgesia. This prospective and double blind study aimed to study the effects of tramadol analgesia associated to dipyrone or ketorolac in the kidney function of patients submitted to LC, using creatinine (Cr), cystatin C, and enzymuria evaluations.

Methods: In the pre- and postoperative (PO) periods, estimated glomerular filtration rates (GFR), obtained from two formulas dependants of blood Cr and one from blood cystatin C values, and tubular enzymuria - alkaline phosphatase (AP), γ-glutamyltransferase (γ-GT) - were determined in patients who underwent LC and analgesia with tramadol and dipyrone (G1, n=63) or tramadol and ketorolac (G2, n=63). In the recovery room (RR), pain and need of rescue analgesia with morphine were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* From 18 to 60 years
* Normal kidney function
* Free consented participation

Exclusion Criteria:

* Renal and hepatic dysfunction
* Prior (one month) use of anti-inflammatory agents

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: adult patients submitted to laparoscopic cholecystectomy and analgesia from tramadol plus ketorolac or dypirone
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2007-02; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yara M Castiglia, MD, PhD, Principal Investigator — Botucatu Medical School
Locations (1):
- UPECLIN, Botucatu, São Paulo, Brazil